CLINICAL TRIAL: NCT07261605
Title: Clinical and Electromyographic Effect of Tui Na Massage Versus Positional Release on Postpartum Neck Dysfunction A Randomized Clinical Trial
Brief Title: Clinical and Electromyographic Effect of Tui Na Massage Versus Positional Release on Postpartum Neck Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, Lecturer of physical therapy department of women health, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PT.BU.EC.20
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Neck Dysfunction
Keywords: electromyographic; Tui-Na massage; positional release; postpartum neck dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- postural correction (Experimental): 20 patients: will receive postural correction exercises program only.
  Interventions: Procedure: postural correction exercises
- Tui NA massage (Experimental): 20 patients: will receive postural correction exercises program. In addition, an experienced therapist will apply the Tui Na massage to the cervical region
  Interventions: Procedure: Tui-Na massage
- Positional release (Experimental): 20 patients: will receive postural correction exercises program. In addition, the therapist put the patient in a comfortable posture for ninety seconds, after which they passively will be moved back to their initial positions
  Interventions: Procedure: positional release

INTERVENTIONS:
Procedure: postural correction exercises — A combination of yoga, stretching, and strengthening exercises may help you to fix or correct your posture over time.
  Maintaining good posture is important for helping you develop strength, flexibility, and balance.
  Arms: postural correction
Procedure: Tui-Na massage — Tuina massage is similar to acupuncture in that it targets specific acupoints, but practitioners use fingers instead of needles to apply pressure to stimulate these points. Tuina massage is often used in combination with acupuncture.
  Arms: Tui NA massage
Procedure: positional release — is a passive manual manipulation method used to alleviate musculoskeletal pain and dysfunction.
  Arms: Positional release

SUMMARY:
To investigate the effects of Tui- Na massage versus Positional release technique on neck pain intensity, neck disability, and electromyographic characteristics of upper trapezius muscle.

DETAILED DESCRIPTION:
Positional release technique

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 20- 40 years
* had post partum cervical pain
* score above 15 in the neck disability index (NDI

Exclusion Criteria:

* Patients with structural, inflammatory, infectious, metabolic, congenital, traumatic spinal disorders and spinal or upper limb surgery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 4 week
  10 cm horizontal line anchored by and it is a line score from zero to ten which 10 score means it is the worse of pain and zero score means the least pain ""no pain"" on the leftand ""worst imaginable pain"" on the right). Patients indicate their pain intensity by marking on the point at the line that reflect their pain
Neck disability index | 4 weeks
  It includes 10 questions of which 7 examine functional activities, 2 ask about symptoms and a question considers concentration.
  Each Patient will circle one of the six options describing the severity of each item (0 5). total score for the questionnaire out of 50. Higher scores represent greater disability.
Electromyography | 4 weeks
  used for measuring upper trapezius normalized Root mean square to indicate muscular activities and median frequence to indicate muscular fatigue. Active electrode will be located 2 cm lateral to the midpoint of a line drawn between C7 spinous process and the posterolateral acromion while the reference one will be located over the C7 spinous process.

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous ishak shehata kelini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No